CLINICAL TRIAL: NCT02277951
Title: Comparison of Four Types of Laryngoscope for Tracheal Intubation During Chest Compressions
Brief Title: Intubation During Resuscitation
Acronym: IDR
Status: Completed | Type: Observational
Sponsor: International Institute of Rescue Research and Education (Other)
Responsible Party: Principal Investigator, Lukasz Szarpak, Lukasz Szarpak, National Institute of Cardiology, Warsaw, Poland
Other Study IDs: InternationalIRRE
Record Dates: First submitted 2014-10-16; First posted 2014-10-29 (Estimated); Last update posted 2014-10-29 (Estimated); Status verified 2014-10

CONDITIONS: Intubation; Cardiopulmonary Resuscitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Participants: The Bonfils Intubation Fibrescope the Video Rigid Flexing Laryngoscope the C-MAC® S Video Laryngoscope the Macintosh Laryngoscope
  Interventions: Device: The Bonfils Intubation Fibrescope; Device: The Video Rigid Flexing Laryngoscope; Device: The C-MAC® S Video Laryngoscope; Device: The Macintosh Laryngoscope

INTERVENTIONS:
Device: The Bonfils Intubation Fibrescope — Effectiveness and time to successful intubation will be measured.
Device: The Video Rigid Flexing Laryngoscope — Effectiveness and time to successful intubation will be measured.
Device: The C-MAC® S Video Laryngoscope — Effectiveness and time to successful intubation will be measured.
Device: The Macintosh Laryngoscope — Effectiveness and time to successful intubation will be measured.

SUMMARY:
The aim of the study was to compare time and success rates of four intubation devices ( in a cardiopulmonary scenario with uninterrupted chest compressions with a standardized manikin model.

The investigators hypothesized that fiberoscope laryngoscopes may improve success rates.

DETAILED DESCRIPTION:
Devices using in study:

The Bonfils Intubation Fibrescope (BONFILS)(KARL STORZ Endovision, Inc., Charlton, MA, USA), The Video Rigid Flexing Laryngoscope (RIFL)( AI Medical Devices, Inc., Williamston, MI, USA), The C-MAC® S Video Laryngoscope Blade Mac#3(C-MAC®S) (KARL STORZ Endovision, Inc., Charlton, MA, USA) The Macintosh Laryngoscope Blade no. 3 (MAC) (LifeLine Medical, Inc., Brooksville, FL, USA).

ELIGIBILITY:
Inclusion Criteria:

* experienced emergency personnel: nurses, paramedics

Exclusion Criteria:

* no experience in out-of-hospital emergency medicine

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Personnel of emergency medical services and hospital emergency units
Sampling Method: Probability Sample
Enrollment: 141 (Actual)
Dates: Start 2014-05; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Time to successful intubation | Subjects complete study in 1 day
  The devices to be compared include (1) The Bonfils Intubation Fibrescope , (2) the Video Rigid Flexing Laryngoscope, (3) the C-MAC® S Video Laryngoscope, (4) the Macintosh Laryngoscope. Successful intubation will be measured in the seconds from insertion of an intubation device to the first manual ventilation of the mannequin's lungs.
Success rate of ETI | Subjects complete study in 1 day
  The devices to be compared include (1) The Bonfils Intubation Fibrescope , (2) the Video Rigid Flexing Laryngoscope, (3) the C-MAC® S Video Laryngoscope, (4) the Macintosh Laryngoscope. Successful intubation will be measured in the seconds from insertion of an intubation device to the first manual ventilation of the mannequin's lungs.